CLINICAL TRIAL: NCT00006721
Title: A Phase III Trial of CHOP Plus Rituximab vs CHOP Plus Iodine-131-Labeled Monoclonal Anti-B1 Antibody (Tositumomab) for Treatment of Newly Diagnosed Follicular Non-Hodgkin's Lymphomas
Brief Title: S0016 Combination Chemotherapy With Monoclonal Antibody Therapy in Newly Diagnosed Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068321; U10CA032102 (NIH); S0016 (Other: SWOG); CALGB-50102 (Other: CALGB); S0016 (Other: ECOG)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Steroids; Vincristine; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (CHOP only) (Active Comparator): Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day
  1. Patients also receive oral prednisone daily on days 1-5. Treatment continues every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. (Arm I closed to accrual as of 12/15/02)
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine
- Arm II (CHOP + rituximab) (Experimental): Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on days 8, 29, 50, 71, 92, and 113. Patients also receive oral prednisone daily on days 8-12, 29-33, 50-54, 71-75, and 113-117 and rituximab IV over 4-6 hours on days 1, 6, 48, 90, 134, and 141.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine
- Arm III (CHOP + tositumomab) (Experimental): Patients receive chemotherapy as in arm I and tositumomab (monoclonal antibody anti-B1) IV over 1 hour followed by iodine I 131 tositumomab IV over 20 minutes on days 134 and 141.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine; Radiation: tositumomab

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: rituxan
  Arms: Arm II (CHOP + rituximab)
Drug: cyclophosphamide — Given IV
  Other Names: cytoxan
Drug: doxorubicin — Given IV
  Other Names: adriamycin
Drug: prednisone — Given orally
  Other Names: steroid
Drug: vincristine — Given IV
  Other Names: oncovin
Radiation: tositumomab — Given IV
  Arms: Arm III (CHOP + tositumomab)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate tumor cells and either kill them or deliver radioactive tumor-killing substances to them without harming normal cells. It is not yet known which monoclonal antibody plus combination chemotherapy regimen is more effective in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is comparing 2 different monoclonal antibodies given together with combination chemotherapy to see how well they work in treating patients with newly-diagnosed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival and overall survival of patients with newly diagnosed follicular non-Hodgkin's lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) with or without either rituximab or iodine I 131 tositumomab (monoclonal antibody anti-B1). (CHOP chemotherapy alone arm closed to accrual as of 12/15/02)
* Compare the response rate of these patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the molecular remission rates of this patient population treated with these regimens.
* Determine the incidence and time to development of human anti-mouse antibody positivity.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to whether microglobulin is greater than upper limit of normal (yes vs no). Patients are randomized to 1 of 3 treatment arms. (Arm I closed to accrual as of 12/15/02)

* Arm I (CHOP only): Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1. Patients also receive oral prednisone daily on days 1-5. Treatment continues every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. (Arm I closed to accrual as of 12/15/02)
* Arm II (CHOP + rituximab): Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on days 8, 29, 50, 71, 92, and 113. Patients also receive oral prednisone daily on days 8-12, 29-33, 50-54, 71-75, and 113-117 and rituximab IV over 4-6 hours on days 1, 6, 48, 90, 134, and 141.
* Arm III (CHOP + tositumomab): Patients receive chemotherapy as in arm I and tositumomab (monoclonal antibody anti-B1) IV over 1 hour followed by iodine I 131 tositumomab IV over 20 minutes on days 134 and 141.

Patients are followed on day 200, at 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 500 patients (250 per treatment arm) will be accrued for this study within 5.5 years. (Arm I closed to accrual as of 12/15/02)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated bulky stage II or stage III or IV follicular non-Hodgkin's lymphoma

  * Grade I-III disease
* Cluster of differentiation antigen 20 (CD20) antigen positive
* Fewer than 5,000/mm^3 circulating lymphoid cells on a white blood cell (WBC) differential count
* Bidimensionally measurable disease
* Bone marrow aspiration and biopsy within the past 42 days
* No clinical evidence of central nervous system (CNS) involvement by lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Granulocyte count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No impaired cardiac status, including:

  * Severe coronary artery disease
  * Cardiomyopathy
  * Congestive heart failure
  * Serious arrhythmia
* Ejection fraction at least lower limit of normal by Multi Gated Acquisition Scan (MUGA) or 2-D echocardiogram for questionable cardiac history

Other:

* No hypersensitivity to iodine
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study participation
* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior monoclonal antibodies for cancer

Chemotherapy:

* No prior chemotherapy for lymphoma

  * Prior prednisone for non-lymphoma related illnesses allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for lymphoma

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2001-03; Primary Completion 2011-09 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Study Chair — Fred Hutchinson Cancer Center; Myron S. Czuczman, MD, Study Chair — Roswell Park Cancer Institute; Sandra J. Horning, MD, Study Chair — Stanford University
Locations (259):
- United States (259):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Sutter Solano Medical Center, Vallejo, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Johnson County Radiation Therapy, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Cancer Center at St. Joseph's Medical Mall, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Radiation Oncology Associates of Kansas City at Northland Radiation Oncology Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Shadman M, Li H, Rimsza L, Leonard JP, Kaminski MS, Braziel RM, Spier CM, Gopal AK, Maloney DG, Cheson BD, Dakhil S, LeBlanc M, Smith SM, Fisher RI, Friedberg JW, Press OW. Continued Excellent Outcomes in Previously Untreated Patients With Follicular Lymphoma After Treatment With CHOP Plus Rituximab or CHOP Plus 131I-Tositumomab: Long-Term Follow-Up of Phase III Randomized Study SWOG-S0016. J Clin Oncol. 2018 Mar 1;36(7):697-703. doi: 10.1200/JCO.2017.74.5083. Epub 2018 Jan 22. PMID 29356608
- [Derived] Press OW, Unger JM, Rimsza LM, Friedberg JW, LeBlanc M, Czuczman MS, Kaminski M, Braziel RM, Spier C, Gopal AK, Maloney DG, Cheson BD, Dakhil SR, Miller TP, Fisher RI. Phase III randomized intergroup trial of CHOP plus rituximab compared with CHOP chemotherapy plus (131)iodine-tositumomab for previously untreated follicular non-Hodgkin lymphoma: SWOG S0016. J Clin Oncol. 2013 Jan 20;31(3):314-20. doi: 10.1200/JCO.2012.42.4101. Epub 2012 Dec 10. PMID 23233710

RESULTS

PARTICIPANT FLOW:
Groups:
- CHOP Only: Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1. Patients also receive oral prednisone daily on days 1-5. Treatment continues every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. (Arm I closed to accrual as of 12/15/02)
- CHOP + Rituximab: Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on days 8, 29, 50, 71, 92, and 113. Patients also receive oral prednisone daily on days 8-12, 29-33, 50-54, 71-75, 92-96 and 113-117 and rituximab IV over 4-6 hours on days 1, 6, 48, 90, 134, and 141
- CHOP + Tositumomab: Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on days 1, 22, 43, 64, 85, and 106. Patients also receive oral prednisone daily on days 1-5, 22-26, 43-47, 64-68, 85-89 and 106-120 and tositumomab (monoclonal antibody anti-B1) IV over 1 hour followed by iodine I 131 tositumomab IV over 20 minutes on days 134 and 141
Period: Overall Study
Arm/Group | CHOP Only | CHOP + Rituximab | CHOP + Tositumomab
Started | 17 | 279 | 275
Eligible | 15 | 267 | 265
Eligible and Began Protocol Therapy | 14 | 267 | 265
Completed | 13 | 254 | 242
Not Completed | 4 | 25 | 33
Not completed — Adverse Event | 0 | 4 | 4
Not completed — Refusal Unrelated to Adverse Event | 1 | 0 | 8
Not completed — Progression/Relapse | 0 | 1 | 2
Not completed — Death | 0 | 1 | 2
Not completed — Other - Not Protocol Specified | 0 | 7 | 7
Not completed — Ineligible | 2 | 12 | 10
Not completed — Eligible but no Treatment Received | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab | CHOP Only | Total
Number analyzed (Participants) | 267 | 265 | 14 | 546
Age, Continuous [Median (Full Range); unit: years] | 54.5 [23.5 to 86.9] | 53.3 [23.6 to 81.8] | 54.5 [32.6 to 75.5] | 54 [23.5 to 86.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 118 | 4 | 247
  Male | 142 | 147 | 10 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 0 | 16
  Not Hispanic or Latino | 232 | 220 | 14 | 466
  Unknown or Not Reported | 29 | 35 | 0 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 5 | 3 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 0 | 21
  White | 241 | 238 | 13 | 492
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 8 | 12 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 2 Years
Description: Measured from time of registration to date of of first observation of progression/relapse, or death due to any cause, or last contact date
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis. The participants in CHOP alone arm were not assessed due to early closure.
Measure: Number; unit: percentage of participants
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 267 | 265
percentage of participants | 76 | 80
Statistical Analysis 1: Comparison: CHOP + Rituximab vs CHOP + Tositumomab; Test type: Superiority or Other; p = 0.11, Regression, Cox; adjusting for the stratification factor (serum beta-2 microglobulin level); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.6 to 1.05] — CHOP + Tositumomab versus CHOP + Rituximab

2. Secondary Outcome: Objective Response (Confirmed and Unconfirmed Complete and Partial Responses)
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: Assessed 200 days and 365 days after initiation of therapy and then every 6 months until death
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 267 | 265
participants | 224 | 223

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal
Time Frame: Patients were assessed for adverse events at end of cycle 1-6 of CHOP or R-CHOP, the end of cycle 1-6 of CHOP and once 2 weeks after the completion of I-131 treatment. For either arm, once 3 months after removal from protocol treatment
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 2.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included
Measure: Number; unit: Participants
Groups:
- CHOP Only: Patients receive cyclophosphamide IV over 15 minutes, doxorubicin IV over 5-20 minutes, and vincristine IV over 5-15 minutes on day 1. Patients also receive oral prednisone daily on days 1-5. Treatment continues every 21 days for up to 6 courses in the abs ence of disease progression or unacceptable toxicity. (Arm I closed to accrual as of 12/15/02)
Arm/Group | CHOP Only | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 13 | 263 | 263
Participants
  ARDS | 0 | 0 | 1
  Abdominal pain/cramping | 0 | 4 | 3
  Allergic reaction | 0 | 9 | 1
  Anemia | 0 | 7 | 8
  Anorexia | 0 | 3 | 2
  Anxiety/agitation | 0 | 1 | 3
  Arrhythmia, NOS | 0 | 1 | 0
  Arthralgia | 0 | 3 | 1
  Arthritis | 0 | 0 | 1
  Ascites (non-malignant) | 0 | 0 | 1
  Ataxia (incoordination) | 0 | 2 | 1
  Bone pain | 0 | 2 | 0
  Cardiac ischemia/infarction | 0 | 1 | 1
  Cardiovascular-other | 0 | 1 | 1
  Cataract | 0 | 1 | 0
  Catheter related infection | 0 | 2 | 0
  Cerebrovascular ischemia | 0 | 1 | 0
  Chest pain,not cardio or pleur | 0 | 4 | 0
  Constipation/bowel obstruction | 1 | 5 | 4
  Cough | 0 | 0 | 1
  Dehydration | 2 | 5 | 1
  Delusions | 0 | 0 | 1
  Depression | 0 | 0 | 2
  Diarrhea without colostomy | 1 | 3 | 3
  Dizziness/light headedness | 0 | 0 | 1
  Double vision | 0 | 1 | 0
  Dyspepsia/heartburn | 0 | 1 | 0
  Dyspnea | 0 | 4 | 4
  Edema | 0 | 0 | 2
  Esophagitis/dysphagia | 0 | 1 | 1
  Fatigue/malaise/lethargy | 0 | 11 | 9
  Febrile neutropenia | 1 | 42 | 26
  Fever without neutropenia | 0 | 1 | 0
  Fever, NOS | 0 | 1 | 0
  Flu-like symptoms-other | 0 | 1 | 0
  Gastric ulcer | 0 | 0 | 1
  Gynecomastia | 0 | 0 | 1
  Headache | 0 | 2 | 1
  Hematologic-other | 0 | 0 | 3
  Hyperglycemia | 0 | 10 | 3
  Hypertension | 0 | 1 | 1
  Hyperuricemia | 0 | 1 | 0
  Hypoalbuminemia | 0 | 1 | 0
  Hypokalemia | 0 | 2 | 2
  Hyponatremia | 0 | 4 | 1
  Hypophosphatemia | 0 | 1 | 0
  Hypotension | 0 | 2 | 1
  Hypoxia | 0 | 1 | 0
  Ileus | 0 | 1 | 0
  Infection w/o 3-4 neutropenia | 0 | 4 | 5
  Infection with 3-4 neutropenia | 0 | 14 | 9
  Infection, unk ANC | 0 | 4 | 3
  Insomnia | 0 | 2 | 1
  Invol. movement/restlessness | 0 | 1 | 0
  Joint,muscle,bone-other | 0 | 0 | 1
  LVEF decrease/CHF | 0 | 1 | 0
  Leukopenia | 4 | 104 | 102
  Lymphopenia | 4 | 64 | 68
  Menses changes | 0 | 2 | 2
  Muscle weakness (not neuro) | 0 | 2 | 3
  Myalgia | 0 | 2 | 3
  Myalgia/arthralgia, NOS | 0 | 2 | 3
  Nausea | 1 | 6 | 10
  Neuro-other | 0 | 0 | 2
  Neuropathic pain | 0 | 1 | 0
  Neutropenia/granulocytopenia | 8 | 127 | 136
  Osteonecrosis | 0 | 0 | 1
  PRBC transfusion | 0 | 2 | 5
  Pain-other | 0 | 2 | 3
  Pancreatitis | 0 | 1 | 0
  Platelet transfusion | 0 | 1 | 7
  Pleural effusions | 0 | 2 | 1
  Pleuritic pain | 0 | 0 | 1
  Pneumonitis/infiltrates | 0 | 0 | 1
  Pruritus | 0 | 1 | 1
  Rash/desquamation | 0 | 1 | 2
  Rectal/perirectal pain | 0 | 0 | 2
  Respiratory infect w/ neutrop | 0 | 3 | 5
  Respiratory infection, unk ANC | 0 | 1 | 2
  SGOT (AST) increase | 0 | 3 | 0
  SGPT (ALT) increase | 0 | 1 | 0
  Second primary | 0 | 0 | 6
  Seizures | 0 | 1 | 0
  Sensory neuropathy | 0 | 10 | 11
  Sinus tachycardia | 0 | 2 | 0
  Skin-other | 0 | 0 | 1
  Speech impairment | 0 | 1 | 0
  Stomatitis/pharyngitis | 0 | 4 | 2
  Supraventricular arrhythmia | 0 | 1 | 0
  Syncope | 0 | 3 | 1
  Thrombocytopenia | 0 | 6 | 47
  Thrombosis/embolism | 0 | 6 | 3
  Tumor lysis syndrome | 0 | 2 | 0
  Urinary frequency/urgency | 0 | 1 | 0
  Urinary tr infection, unk ANC | 0 | 1 | 0
  Vaginal bleeding | 0 | 0 | 1
  Voice change/stridor/larynx | 0 | 0 | 1
  Vomiting | 1 | 4 | 10
  Weakness (motor neuropathy) | 1 | 4 | 4
  Weight loss | 0 | 0 | 2

4. Primary Outcome: Progression-free Survival at 5 Years
Description: as for outcome 1
Time Frame: 0-5 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 267 | 265
percentage of participants | 60 | 66

5. Primary Outcome: Overall Survival at 2 Years
Description: Measured from date of registration to date of death due to any cause
Time Frame: 0-2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 267 | 265
percentage of participants | 97 | 93
Statistical Analysis 1: Comparison: CHOP + Rituximab vs CHOP + Tositumomab; Test type: Superiority or Other; p = 0.08, Regression, Cox; adjusting for the stratification factor (serum beta-2 microglobulin level); Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.95 to 2.54] — CHOP + Tositumomab versus CHOP + Rituximab

6. Primary Outcome: Overall Survival at 5 Years
Description: Measured from date of registration to date of death due to any cause
Time Frame: 0-5 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CHOP + Rituximab | CHOP + Tositumomab
Number analyzed (Participants) | 267 | 265
percentage of participants | 92 | 86

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events at end of cycle 1-6 of CHOP or R-CHOP, the end of cycle 1-6 of CHOP and once 2 weeks after the completion of I-131 treatment. For either arm, once 3 months after removal from protocol treatment
Arm/Group | CHOP Only | CHOP + Rituximab | CHOP + Tositumomab
Serious Adverse Events (participants affected / at risk) | 0/13 | 3/263 | 16/263
Other Adverse Events (participants affected / at risk) | 13/13 | 262/263 | 261/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP Only (N=13) | CHOP + Rituximab (N=263) | CHOP + Tositumomab (N=263)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Hematologic-other (Blood and lymphatic system disorders) | 0 | 0 | 3
Platelet transfusion (Blood and lymphatic system disorders) | 0 | 0 | 1
LVEF decrease/CHF (Cardiac disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Infection w/o 3-4 neutropenia (Infections and infestations) | 0 | 0 | 2
Respiratory infect w/ neutrop (Infections and infestations) | 0 | 0 | 1
Neutropenia/granulocytopenia (Investigations) | 0 | 0 | 1
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6
Cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP Only (N=13) | CHOP + Rituximab (N=263) | CHOP + Tositumomab (N=263)
Anemia (Blood and lymphatic system disorders) | 5 | 177 | 192
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 42 | 24
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal pain/cramping (Gastrointestinal disorders) | 2 | 61 | 47
Constipation/bowel obstruction (Gastrointestinal disorders) | 4 | 106 | 99
Diarrhea without colostomy (Gastrointestinal disorders) | 3 | 57 | 61
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 38 | 40
Esophagitis/dysphagia (Gastrointestinal disorders) | 1 | 17 | 0
GI-other (Gastrointestinal disorders) | 0 | 16 | 0
Nausea (Gastrointestinal disorders) | 6 | 149 | 173
Stomatitis/pharyngitis (Gastrointestinal disorders) | 5 | 90 | 84
Vomiting (Gastrointestinal disorders) | 5 | 56 | 83
Edema (General disorders) | 2 | 45 | 33
Fatigue/malaise/lethargy (General disorders) | 7 | 207 | 198
Fever without neutropenia (General disorders) | 0 | 35 | 24
Fever, NOS (General disorders) | 1 | 0 | 0
Pain-other (General disorders) | 0 | 57 | 42
Rigors/chills (General disorders) | 2 | 65 | 29
Sweating (General disorders) | 0 | 56 | 33
Allergic reaction (Immune system disorders) | 1 | 49 | 0
Infection w/o 3-4 neutropenia (Infections and infestations) | 0 | 42 | 39
Infection with 3-4 neutropenia (Infections and infestations) | 0 | 17 | 0
Respiratory infect w/o neutrop (Infections and infestations) | 0 | 15 | 14
Alkaline phosphatase increase (Investigations) | 0 | 22 | 15
Creatinine increase (Investigations) | 0 | 17 | 15
Leukopenia (Investigations) | 11 | 187 | 205
Lymphopenia (Investigations) | 7 | 145 | 155
Neutropenia/granulocytopenia (Investigations) | 10 | 174 | 187
SGOT (AST) increase (Investigations) | 2 | 41 | 45
SGPT (ALT) increase (Investigations) | 0 | 26 | 41
Thrombocytopenia (Investigations) | 3 | 77 | 140
Weight loss (Investigations) | 0 | 26 | 31
Anorexia (Metabolism and nutrition disorders) | 3 | 63 | 59
Dehydration (Metabolism and nutrition disorders) | 2 | 21 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 79 | 77
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 22 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 24 | 15
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 15
Hypokalemia (Metabolism and nutrition disorders) | 0 | 16 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 22 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 37 | 41
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 16 | 0
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 0 | 20 | 0
Joint,muscle,bone-other (Musculoskeletal and connective tissue disorders) | 0 | 14 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 63 | 57
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 0 | 25 | 40
Dizziness/light headedness (Nervous system disorders) | 1 | 22 | 20
Headache (Nervous system disorders) | 3 | 61 | 52
Sensory neuropathy (Nervous system disorders) | 7 | 120 | 119
Taste disturbance (Nervous system disorders) | 0 | 29 | 30
Weakness (motor neuropathy) (Nervous system disorders) | 2 | 27 | 22
Anxiety/agitation (Psychiatric disorders) | 1 | 34 | 38
Depression (Psychiatric disorders) | 2 | 20 | 31
Insomnia (Psychiatric disorders) | 2 | 60 | 59
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 16 | 21
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 23 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 71 | 43
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 52 | 44
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 176 | 151
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pigmentation changes/yellowing (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 17 | 16
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 37 | 44
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 0 | 16
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 14 | 0
Hypotension (Vascular disorders) | 1 | 16 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No